The First Affiliated Hospital of Gannan Medical University, Department of Rehabilitation Medicine

Clinical Research Recruitment Announcement for Patients with Disorders of Consciousness after Craniocerebral Injury

Ethics Approval Number: LLSL-2022053105

Date: February 2022

The First Affiliated Hospital of Gannan Medical University,

Department of Rehabilitation Medicine

Clinical Research Recruitment Announcement for Patients with
Disorders of Consciousness after Craniocerebral Injury
Dear Patients and Family Members:

Our hospital is currently conducting a clinical research study titled "Median Nerve Electrical Stimulation Combined with Auricular Point Acupuncture for Disorders of Consciousness after Craniocerebral Injury." We are now openly recruiting eligible patients. The details are as follows:

## I. Recruitment Criteria

Patients with disorders of consciousness after brain injury, with a Glasgow Coma Scale (GCS) score between 4 and 8, and a disease duration of  $\leq 10$  days.

Stable vital signs, without severe organ failure, history of epilepsy, or previous craniocerebral injury.

Family members are informed and provide consent, and are willing to cooperate with the treatment.

## II. Research Content

Eligible participants will be randomly divided into two groups. They will receive either conventional treatment combined with median nerve electrical stimulation, or conventional treatment combined with median nerve electrical stimulation and

auricular point acupuncture. The treatment period will last for

8 weeks.

III. Participant Rights

Relevant examinations and treatments during the study will

be provided free of charge.

A professional medical team will monitor the patient's

condition throughout the study.

Participants may withdraw from the study at any time without

affecting their routine treatment.

IV. Registration Method

Contact Person: Liao Jinghai

Phone: 15297770567

Address: Rehabilitation Therapy Room, 2nd Floor, North

Inpaient Building

Ethics Approval Number: LLSL-2022053105

This study complies with medical ethics requirements and

strictly protects participants' privacy.

Department of Rehabilitation Medicine

February 2022